CLINICAL TRIAL: NCT04775264
Title: Safety and Feasibility of Atrial Deganglionation as Adjunctive Therapy for Atrial Fibrillation
Brief Title: Safety and Feasibility of Atrial Deganglionation as Adjunctive Therapy for AF
Acronym: Neural-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atrian Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulsed Electric Field Energy Ablation (Experimental): Ablation of ganglionated plexi (GP) structures on the epicardial surface of the heart delivered as a concomitant procedure during open heart surgery.
  Interventions: Procedure: Pulsed Electric Field Ablation

INTERVENTIONS:
Procedure: Pulsed Electric Field Ablation — Catheter ablation of Ganglionated Plexi (GP) structures on the epicardial surface of the heart during cardiothoracic surgery

SUMMARY:
A prospective, single arm, multi-center exploratory study of safety and feasibility in the treatment of patients undergoing cardiothoracic surgery.

DETAILED DESCRIPTION:
To assess the safety and feasibility of electroporation/Pulsed Electric Field (PEF) as a technology to achieve selective GP ablation. This treatment will be performed on 30 patients undergoing cardiothoracic surgery. Primary feasibility endpoint will be demonstration of ability to access and deliver Pulsed Electric Field energy to all of the targeted ablation sites.

ELIGIBILITY:
Inclusion Criteria:

* Age is between 18 and 70 years.
* Scheduled for open-chest cardiothoracic surgery, for coronary artery bypass grafting.
* Legally competent and willing to sign the informed consent.
* Life expectancy of at least 2 years.

Exclusion Criteria:

* • Previous cardiac surgery.

  * Prior pericardial interventions.
  * Prior pulmonary vein isolation (PVI).
  * Previous or existing pericarditis.
  * Persistent or long-standing persistent atrial fibrillation.
  * Indication for surgical ablation or PVI for atrial fibrillation.
  * Indication for concomitant surgical valve repair or replacement.
  * Indication for concomitant left atrial appendage (LAA) ligation or excision.
  * History of previous radiation therapy on the thorax.
  * History of previous thoracotomy.
  * Prior electrical or mechanical isolation of the Left Atrial Appendage (LAA).
  * The presence of LAA occlusion devices, coronary stents, prosthetic heart valves, pacemakers or implantable cardioverter defibrillators (ICDs).
  * Myocardial infarction within the previous 2 months.
  * NYHA (New York Heart Association) Class IV heart failure symptoms.
  * Left ventricular ejection fraction (LVEF) < 40%, measured by transthoracic echocardiography (TTE).
  * Left atrial (LA) diameter > 5.0 cm, measured by transthoracic echocardiography (TTE).
  * The presence of left atrial thrombus when examined by transoesophageal echocardiography (TEE).
  * The presence of AF attributable to non-cardiovascular causes such as thyroid disease, electrolyte imbalance/dehydration or other reversible causes.
  * Active infection or sepsis as evidenced by increased white blood cell count, elevated CRP (C-Reactive Protein) or temperature > 38.5°C.
  * Known or documented carotid stenosis > 80%
  * Stroke or transient ischemic attack within the previous 6 months.
  * Known or documented epilepsy.
  * Pregnancy or child-bearing potential without adequate contraception.
  * Circumstances that prevent follow-ups.
  * Drug abuse.
  * Patients cannot be enrolled in another clinical study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry O'Brien, PhD, Study Chair — AtriAN Medical
Locations (2):
- Na Homolce Hospital, Prague, Czechia
- Tbilisi Heart & Vascular Clinic, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Musikantow DR, Reddy VY, Skalsky I, Shaburishvili T, van Zyl M, O'Brien B, Coffey K, Reilly J, Neuzil P, Asirvatham S, de Groot JR. Targeted ablation of epicardial ganglionated plexi during cardiac surgery with pulsed field electroporation (NEURAL AF). J Interv Card Electrophysiol. 2025 Mar;68(2):467-474. doi: 10.1007/s10840-023-01615-8. Epub 2023 Aug 10. PMID 37561246

RESULTS

PARTICIPANT FLOW:
Groups:
- Pulsed Electric Field Ablation of Ganglionated Plexi: Pulsed Electric Field Ablation: Catheter ablation of ganglionated plexi structures on the epicardial surface of the heart during cardiothoracic surgery.
Period: Overall Study
Arm/Group | Pulsed Electric Field Ablation of Ganglionated Plexi
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pulsed Electric Field Ablation of Ganglionated Plexi
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Czechia | 8
  Georgia | 16
Body Mass Index [Mean (Standard Deviation); unit: Kg/m˄2] | 29.4 (4.4)
Left Atrial Diameter [Mean (Standard Deviation); unit: cm] | 3.7 (0.4)
Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: % (of total left ventricle volume)] | 49.7 (7.4)
Paroxysmal AF History [Count of Participants; unit: Participants] | 3
Coronary Artery Disease [Count of Participants; unit: Participants] | 22
Prior Myocardial Infarction [Count of Participants; unit: Participants] | 2
Hypertension [Count of Participants; unit: Participants] | 23
Diabetes [Count of Participants; unit: Participants] | 9
Stroke or TIA (Transient Ischemic Attack) [Count of Participants; unit: Participants] | 0
Beta Blockers [Count of Participants; unit: Participants] | 19
Class I or III anti-arrhythmic [Count of Participants; unit: Participants] | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device-related Primary Safety Adverse Events
Description: Primary Safety Adverse Events include:
  1. Atrial perforation or excessive bleeding (excessive bleeding is defined as bleeding which requires any blood transfusion).
  2. Pericarditis
  3. Pericardial effusion
  4. Cardiac tamponade (if either surgical or percutaneous drainage is required).
  5. Constrictive pericarditis, requiring re-operation.
  6. Newly developed sinus node dysfunction.
  7. Newly developed first, second or third degree atrioventricular (AV) block
  8. Vasovagal reactions during hospital stay
  9. Ventricular fibrillation
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsed Electric Field Ablation of Ganglionated Plexi
Number analyzed (Participants) | 24
Participants | 0

2. Primary Outcome: Number of Participants in Which Pulsed Electric Field Was Successfully Delivered to All Target Sites on the Epicardial Surface of the Heart.
Description: Confirmation of catheter access and delivery of pulsed electric field energy to each of the targeted ablation sites on the epicardial surface of the heart.
Time Frame: Intraprocedural - during the ablation procedure. Within 1 hour of sternotomy.
Measure: Count of Participants; unit: Participants
Arm/Group | Pulsed Electric Field Ablation of Ganglionated Plexi
Number analyzed (Participants) | 24
Participants | 24

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Pulsed Electric Field Ablation of Ganglionated Plexi
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 3/24
Other Adverse Events (participants affected / at risk) | 5/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Electric Field Ablation of Ganglionated Plexi (N=24)
Post-operative Atrial Fibrillation (Cardiac disorders) | 2 (2) — Post-operative Atrial Fibrillation requiring electrical cardioversion
Pulmonary Embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulsed Electric Field Ablation of Ganglionated Plexi (N=24)
Intra-procedural Hypotension and Atrial Fibrillation (Cardiac disorders) | 1 (1) — Hypotension and Atrial Fibrillation during delivery of ablation energy
Intra-procedural Atrial Fibrillation (Cardiac disorders) | 1 (1) — Atrial Fibrillation during delivery of ablation energy
Atrial Fibrillation (Cardiac disorders) | 1 (1) — Atrial Fibrillation during index Coronary Artery Bypass Grafting procedure
Post-operative Atrial Fibrillation (Cardiac disorders) | 4 (5) — Post-operative Atrial Fibrillation resolved with chemical cardioversion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT04775264/Prot_SAP_000.pdf